CLINICAL TRIAL: NCT04400539
Title: Intrapleural Photodynamic Therapy by Video-Assisted Thoracoscopy Followed by Anti-PD-1 NIVOLUMAB in Patients With Malignant Pleural Mesothelioma - a Pilot Study
Brief Title: The IMmunotherapy Pleural 5-ALA PDT
Acronym: IMPALA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: INSERM U1189 ONCOTHAI (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019_41; 2019-003003-35 (EudraCT Number)
Record Dates: First submitted 2020-05-20; First posted 2020-05-22 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Mesotheliomas Pleural; Malignant Pleural Mesothelioma
Keywords: Immunotherapy; anti-PD-1; Photodynamic Therapy
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — Thoracic Surgery, Video-Assisted; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Malignant Pleural Mesothelioma patients (Experimental)
  Interventions: Device: intrapleural photodynamic therapy with videothoracoscopy; Drug: Nivolumab Injection

INTERVENTIONS:
Device: intrapleural photodynamic therapy with videothoracoscopy — MPM patients will be first administrated 20 mg/kg of oral photosensitizer, 5-Aminolevulinic Acid (5-ALA) {Gliolan®}, 4 to 6 hours prior undergoing thoracoscopy (VATS). During VATS procedure, after a qualitative control of the fluorescence of tumor lesions and some guided pleural tumor biopsies, the pleural cavity will be illuminated using a flexible probe and laser source at a specific wavelength for 5-ALA (400-500 nm; 25 J/cm2) during 15 minutes (6 fractions of 2.5 minutes separated by 5 pauses of 2 minutes each to improve tissue oxygenation for the PDT reaction). An IPC device (but no talc) will be inserted and used for pleurodesis and may permit to collect further pleural effusion samples. As 5-ALA has a short half-life and thus does not need extensive precautions to avoid patient photosensitivity, the patient would not stay longer than a standard procedure (about 2-3 days in the hospital)
Drug: Nivolumab Injection — Seven to 10 days after VATS, patients will start to be treated by Nivolumab 240mg IV every 2 weeks till progression (CT-scan reassessment every 8 cycles), unacceptable toxicity, or maximum 2 years.
  Other Names: adjuvant immunotherapy with anti-PD-1 Nivolumab antibodies

SUMMARY:
Pilot study of the feasibility of an innovative multimodal treatment combining intrapleural photodynamic therapy with videothoracoscopy followed by adjuvant immunotherapy with anti-PD-1 Nivolumab antibodies in patients with malignant pleural mesothelioma

ELIGIBILITY:
Inclusion Criteria:

* ECOG Performance status (PS) 0-1 (WHO)
* Unresectable Malignant Pleural Mesothelioma
* suffering from unresectable MPM (n=20), relapsing after one or 2 lines of treatment with platinum-based doublet of chemotherapy (including pemetrexed) [Note: MPM patients having contra-indications for, or refusing chemotherapy may also be recruited], and candidate for palliative pleural procedure (i.e. thoracoscopy for pleurodesis by talc or by insertion of indwelled pleural catheter, IPC)
* Documented progression after previous 1 or 2 lines of chemotherapy including Platinum/Pemetrexed chemotherapy*
* Measurable disease according to modified RECIST 1.1. for MPM
* Malignant pleural lesion assessed to be accessible by local PDT treatment during thoracoscopy, as validated by expert MTB ("MESOCLIN", Lille, France)
* Histological diagnosis confirmed by national expert pathology panel ("MESOPATH" - Institut Léon Bérard, Lyon, France)
* Weight loss <10%
* available tumor tissue (archival or fresh)
* obtention of an informed written consent before any specific procedure of the study
* Decision to treat the patient within this clinical trial taken during MPM dedicated multidisciplinary board (RCP MESOCLIN in France )
* Patient affiliated to and covered by social security for standard care
* Women of child-bearing potential must use a highly effective method of contraception for 28 days prior to the first dose of investigational product, and must agree to continue using such precautions for 5 months after the final dose of investigational product
* Women of child-bearing potential must have a negative pregnancy test within 24h before administration of investigational product
* First line patients may also be recruited if they declined or if they have contra-indications for chemotherapy.

Exclusion Criteria:

* lack of informed written consent; or refusal to sign or to participate
* Pregnant, breastfeeding patients, and female patients of childbearing potential who are unwilling or unable to use a highly effective method of contraception as outlined in the protocol for the duration of the study and for at least 5 months after the last dose of nivolumab
* Male patients who are unwilling or unable to use contraception methods for the duration of the study and for at least 7 months after the last dose of nivolumab
* a previous treatment by anti-PD-1 or anti-PD-L1 antibodies for their cancer or any other cancer in the last 5 years
* hypersensitivity to Nivolumab (anti-PD-1 antibodies)
* contra-indications for 5-ALA or PDT
* contra-indications for thoracoscopy (VATS)
* any other comorbidity precluding the feasibility of the therapeutic protocol: uncontrolled cardiac failure, pulmonary hypertension, liver or kidney severe dysfunction (creatinin clearance <60 ml/min), uncontrolled infection, or other disease according to the investigator
* other cancer treated within 5 years before inclusion except baso-cellular skin carcinoma or cervical / bladder in situ carcinoma
* inability to receive study information and to give informed consent
* patient unable to have a clinical follow-up due to psychological, familial, social or geographical reasons
* legal incapacity (people in jail), or under supervision (i.e. guardianship or curatorship)
* treatment with experimental drug within 30 days before the start of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-05-09 (Actual); Primary Completion 2026-05-09 (Estimated); Study Completion 2026-05-09 (Estimated)

PRIMARY OUTCOMES:
the proportion of patients having the full multimodal treatment | through study completion, an average of 24 months
  the proportion of patients having the full multimodal treatment (target: 70% minimum of total patients,14 out of 20 patients) without inacceptable and unexpected toxicity (grade≥3) according National Cancer Institute (NCI) criteria, reviewed by an Independent Survey Committee.

SECONDARY OUTCOMES:
objective response rate (ORR) according to modified RECIST 1.1 criteria for mesothelioma for pleural lesions; RECIST 1.1 for all other targets | through study completion, an average of 24 months
Kaplan Meier curve for overall survival (mOS) | through study completion, an average of 24 months
Kaplan Meier curve for progression free survival (mPFS) | through study completion, an average of 24 months
quality of life (QoL) of patients by dedicated EORTC QLQ C30 (or LCSS-30) questionnaire | At baseline and
  The Quality of life questionnaire (QLQ-C30) contains 29 items dealing with fatigue, pain, nausea and vomiting, general condition and social, emotional and cognitive functions. It is currently used in many clinical trials in oncology
evaluation of chest pain using visual scale. | through study completion, an average of 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud Scherpereel, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Institut Coeur-Poumon, CHU, Lille, France